CLINICAL TRIAL: NCT02553213
Title: Early Changes of Diabetes Parameters After Obesity Therapy
Acronym: ECODO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Hohenheim (Other)
Collaborators: University Hospital Tuebingen (Other); Karl-Olga-Krankenhaus Stuttgart (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Studie_ECODO
Record Dates: First submitted 2015-09-04; First posted 2015-09-17 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Bariatric Surgery Candidate
MeSH Terms: interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LSG group (Experimental): Laparoscopic sleeve gastrectomy
  Interventions: Other: Laparoscopic sleeve gastrectomy; Other: easy digestible diet
- LRYGB group (Experimental): Laparoscopic Roux-en-Y gastric bypass
  Interventions: Other: Laparoscopic Roux-en-Y gastric bypass; Other: easy digestible diet
- Control group (Other): Caloric restriction
  Interventions: Other: Caloric restriction diet

INTERVENTIONS:
Other: Laparoscopic sleeve gastrectomy — The surgical procedure and aftercare is indicated and performed according to the routine clinical setting of the Hospital. Patients stay 5 days stationary after surgical treatment. They receive a defined easy digestible diet, starting with liquid and mash food.
  Arms: LSG group
Other: Laparoscopic Roux-en-Y gastric bypass — The surgical procedure and aftercare is indicated and performed according to the routine clinical setting of the Hospital. Patients stay 5 days stationary after surgical treatment. They receive a defined easy digestible diet, starting with liquid and mash food.
  Arms: LRYGB group
Other: Caloric restriction diet — Patients of the control group do not undergo surgical treatment. They undergo a caloric restriction diet for 5 days. This diet is adapted to the postoperative diet of the patients included in the two other groups.
  Arms: Control group
Other: easy digestible diet
  Arms: LRYGB group; LSG group

SUMMARY:
The aim of the study is to investigate, if bariatric surgery or the related caloric restriction causes the significant improvement of glucose metabolism, which has been found in bariatric patients.

DETAILED DESCRIPTION:
Previous studies have shown, that laparoscopic Roux-en-Y gastric bypass (LRYGB), and also laparoscopic sleeve gastrectomy (LSG) leed to a significant improvement of glucose metabolism and in many cases to a complete remission of diabetes type II in obese patients. It is still unclear which mechanisms underlie these changes. Since the positive effects of bariatric surgery have been investigated within few days after surgical intervention, before significant weight loss has been achieved, the caloric restriction has been discussed as a possible mechanism.

The aim of the study is to investigate, if bariatric surgery or the related caloric restriction causes the significant improvement of glucose metabolism, which has been found in bariatric patients. Therefore, the investigator will examine obese patients with diabetes type II or impaired glucose metabolism regarding possible metabolic changes within few days after bariatric surgery (LSG or LRYGB) or caloric restriction only.

Group I: Patients undergoing LSG; Group II: Patients undergoing LRYGB; Group III (Control group): Patients undergoing caloric restriction;

Dietetic, anthropometric, metabolic and hormonal parameters will be measured. Primary outcome marker is the insulin sensitivity according to Matsuda (MISI).

The project is a prospective, controlled study. Study examinations will be performed before intervention, and one, two, three, four and five days after (start of) intervention, as well after one month.

ELIGIBILITY:
Inclusion Criteria:

* BMI (Body Mass Index) ≥ 35 kg/m2
* Clinical diagnosis of type II diabetes or impaired glucose metabolism (Prediabetes: HbA1c > 5,7%, fasting glucose in capillary blood > 110 mg/dl - diagnosed by blood glucose test at the first study examination)
* Regarding the patients of the surgical groups: Indication to surgical therapy of obesity (laparoscopic sleeve gastrectomy or Roux-en-Y gastric bypass). The indication to surgery is independent of the study. The surgeon decides about that in the clinical routine according to the German S3 guideline.
* Written consent to participate int he study

Exclusion Criteria:

* Medication use which affects glucose metabolism, except for diabetes medication (for example: glucocorticoids)
* Insulin need >1,0 IU/kg/d
* Experimental diabetes medication within the last three months
* Pregnancy
* Gastrointestinal diseases
* Uncontrolled hypo- or hyperthyroidism
* Status after bariatric or other gastrointestinal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-05 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change of insulin | Within 5 days after surgery or 5 days after start of caloric restriction
  Blood insulin is measured during a Mixed Meal Tolerance Test (MMTT). It is used to calculate the Homeostasis Model Assessment (HOMA) and Matsuda Insulin Sensitivity Index
Change of blood glucose | Within 5 days after surgery or 5 days after start of caloric restriction
  Blood glucose is measured during a Mixed Meal Tolerance Test (MMTT). It is used to calculate the Homeostasis Model Assessment (HOMA) and Matsuda Insulin Sensitivity Index

OTHER OUTCOMES:
Changes regarding markers of glucose metabolism | Within 5 days after surgery or 5 days after start of caloric restriction
  HbA1c, C-Peptid, insulin and fasting glucose
Changes of body weight | Within 5 days after surgery or 5 days after start of caloric restriction
Changes of blood lipids | Within 5 days after surgery or 5 days after start of caloric restriction
  High density lipoprotein, low density lipoprotein, triglycerides, free fatty acids
Changes concerning the intake of calories and nutrients | Within 5 days after surgery or 5 days after start of caloric restriction
  Measured by using nutritional protocols
Changes of gastrointestinal hormones | Within 5 days after surgery or 5 days after start of caloric restriction
  Glucagon-like peptide-1, Ghrelin, Glucose-dependent insulinotropic peptide
Changes of adiponectin | Within 5 days after surgery or 5 days after start of caloric restriction
Changes of bile acids | Within 5 days after surgery or 5 days after start of caloric restriction
Changes of gut microbiota composition | Within 5 days after surgery or 5 days after start of caloric restriction
Changes of body height | Within 5 days after surgery or 5 days after start of caloric restriction
Changes of body composition | Within 5 days after surgery or 5 days after start of caloric restriction
  measured by Body Impedance Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C. Bischoff, Prof., Study Chair — Department of Nutritional Medicine, University of Hohenheim, Stuttgart, Germany; Alfred Königsrainer, Prof., Study Director — Department of General, Visceral, and Transplant Surgery, University Hospital Tübingen, Germany
Locations (1):
- University of Hohenheim, Stuttgart, Germany